CLINICAL TRIAL: NCT00543790
Title: A Randomized, Placebo-Controlled, Double-Blind, Sponsor-Unblinded, Multiple-Dose Study Of The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of PRA-027 Administered Orally To Cycling Or Postmenopausal Women
Brief Title: Study Evaluating PRA-027 Multiple Ascending Doses In Cycling And Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3208A1-1001; B2531001
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Uterine Leiomyomata (Fibroids)
MeSH Terms: conditions — Myofibroma; Leiomyoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PRA-027

INTERVENTIONS:
Drug: PRA-027 — PRA-027 capsules; cohort-specific doses or 40, 120, 240 or 500 mg; 1 dose daily for 28 days

SUMMARY:
This is the first multiple-dose study in humans with PRA-027. This study will provide an assessment of the safety, tolerability, pharmacokinetics (how the drug is absorbed, metabolized and excreted by the body) and pharmacodynamics (a measure of whether the drug is active in the body) of PRA-027 after administration of 28 days of oral doses in women of childbearing potential (cycling) or postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - All Women

* Healthy, nonsmoker or smoker of fewer than 10 cigarettes (half a pack) per day and able to abstain from tobacco throughout all times when in the clinical facility.

Inclusion Criteria - Cycling Women

* Aged 18 to 45 years, must not be breastfeeding, pregnant, or have a recent (within 90 days before pretreatment period day 1) history of pregnancy, with a history of regular menstrual cycles (21 to 35 days in duration).

Inclusion Criteria - Postmenopausal Women

* Aged 35 to 65 years, menopause may be natural or due to surgery, natural amenorrhea must have begun by age of 55 years and have initiated at least 6 months before study day 1.

Exclusion Criteria:

* Women with hysterectomy or complex or simple ovarian cysts greater than 3 cm in diameter.
* History of drug abuse (within 6 months) or alcoholism (within 12 months).
* History of female infertility.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of ascending, multiple, oral doses of PRA-027 in cycling and postmenopausal women. | 28 days

SECONDARY OUTCOMES:
To provide the PK and PD profile of multiple oral doses of PRA-027 in cycling and postmenopausal women. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Miami, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3208A1-1001&StudyName=Study%20Evaluating%20PRA-027%20Multiple%20Ascending%20Doses%20In%20Cycling%20And%20Postmenopausal%20Women